CLINICAL TRIAL: NCT00786006
Title: Randomized Phase II Trial of FOLFIRI3 vs. FOLFOX in Gemcitabine-refractory Advanced Pancreatic Cancer
Brief Title: Randomized Phase II Study of FOLFOX Versus FOLFIRI.3 in Gemcitabine-refractory Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC_P_01
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; gemcitabine; oxaliplatin; irinotecan; fluorouracil; Failure to gemcitabine chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): FOLFIRI.3
  Interventions: Drug: FOLFIRI.3
- Arm 2 (Active Comparator): FOLFOX
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: FOLFIRI.3 — FOLFIRI.3: Irinotecan 70 mg/m2 (over 60 min) on D1, LV 400 mg/m2 (over 2h) D1, 5-FU 2000 mg/m2 (over 46 hours) from D1, then irinotecan 70 mg/m2(over 60 min) at the end of the 5-FU infusion
  Arms: Arm 1
Drug: FOLFOX — FOLFOX: oxaliplatin 85 mg/m2 (over 120 min) on D1, LV 400 mg/m2 (over 2hour) on D1, 5-FU 400 mg/m2 IVP on D1, 5-FU 2,000 mg/m2 (over 46 hours)
  Arms: Arm 2

SUMMARY:
The investigators are to evaluate the efficacy and safety of FOLFOX or FOLFIRI.3 combination chemotherapy as second-line salvage chemotherapy in patients with advanced pancreatic carcinoma.

DETAILED DESCRIPTION:
Given the poor response rate, usually less than 20% in gemcitabine-based doublet in the first-line setting for advanced pancreatic cancer, an additional problem in the therapeutic management of this common malignant disease constitutes the need for effective treatment alternatives in patients failing gemcitabine-based chemotherapy. To date, few studies have assessed second-line chemotherapy primarily due to the poor prognosis, and the limited life expectancy in advanced pancreatic cancer after failure first-line chemotherapy, and there has been no established second-line treatment for pancreatic cancer after failure to gemcitabine.

1. Oxaliplatin combination with 5-FU (FOLFOX)

   Oxaliplatin, diaminocyclohexane-platinum, is an alkylating agent inhibiting DNA replication by forming adducts between two adjacent guanines or guanine and adenine molecules. With regard to the inhibition of DNA synthesis, the adducts of oxaliplatin appear to be more effective than cisplatin adducts. Synergism between oxaliplatin and 5-FU has been demonstrated in vitro, and in vivo. Combination of oxaliplatin and 5-FU has proven effective as first- or second-line treatment for advanced colorectal cancer. After being extensively developed as a treatment for colorectal cancer, the role for oxaliplatin in upper gastrointestinal malignancies including pancreatic cancer is an emerging area of investigation. In preclinical studies, oxaliplatin has cytotoxic activity against pancreatic cancer cell lines. When used as single agent as first-line treatment or as second-line treatment after failure to gemcitabine-based chemotherapy, oxaliplatin has minimal activity against pancreatic cancer. However, when it is used with 5-FU, it produced 10% objective response rate with a 21% of clinical benefit response with minimal toxicities in chemotherapy-naïve patients. In phase II studies as second-line treatment, oxaliplatin with 5-FU is well tolerated and produced a objective response rate of 23.3% with additional 30.0% of patients achieving stable disease. Furthermore, recently Oettle et al. reported that weekly infusional 5FU/LV with oxaliplatin prolongs survival and improves quality of life in advanced pancreatic cancer after gemcitabine failure compared with best supportive care alone.
2. Irinotecan combination with 5-FU (FOLFIRI.3)

Irinotecan has a strong growth-inhibiting effect on cultured pancreatic adenocarcinoma cells. It is also highly active on pancreatic tumor cells in culture and in xenograft models. Irinotecan monotherapy has been tested in patients with previously untreated pancreatic cancer, yielding response rates of 9-27%. In vitro studies indicate that synergism between irinotecan and 5-FU is sequence dependent, cytotoxicity is being stronger when irinotecan is administered before 5-FU. Recently, French study group reported that FOLFIRI.3 regimen, comprising of irinotecan D1 and D3 with 5-FU for 2 days from D2, has promising activity in chemotherapy-naïve and pretreated patients with advanced pancreatic cancer. The confirmed response rate was 37.5% with a median progression-free survival of 5.6 months. The study also suggested no cross-resistance between gemcitabine and FOLFIRI.3.

The investigators are to evaluate the efficacy and safety of FOLFOX or FOLFIRI.3 combination chemotherapy as second-line salvage chemotherapy in patients with advanced pancreatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven pancreatic adenocarcinoma
2. Age 18 year or older
3. ECOG performance status of 2 or lower
4. Documented disease progression while receiving or within 6 months after discontinuing gemcitabine-based first-line or adjuvant chemotherapy
5. Adequate bone marrow function A. WBCs > 4,000/µL, absolute neutrophil count [ANC]>1,500/µL B. Hemoglobin >9.0 g/dL C. Platelets > 100,000/µL
6. Adequate kidney function (creatinine<1.5 mg/dL)
7. Adequate liver function (bilirubin<1.5 mg/dL [< 2.5 mg/dL for obstructive jaundice with adequately decompressed bile duct obstruction], transaminases levels<3 times the upper normal limit, and serum albumin of >2.5 mg/dL)
8. No serious other medical condition that would preclude treatment

Exclusion Criteria:

1. Other tumor type than adenocarcinoma
2. Evidence of GI bleeding or GI obstruction
3. Presence or history of CNS metastasis
4. Axial skeletal radiotherapy within 6 months
5. Neuropathy grade 2 or worse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | Every 6 weeks

SECONDARY OUTCOMES:
Response rate | Every 6 weeks
Overall survival | every 6 weeks during treatment and every 2 months after off-treatment
Safety | Every 2 weeks
  NCI CTCAE v.3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD, PhD, Study Chair — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Result] Yoo C, Hwang JY, Kim JE, Kim TW, Lee JS, Park DH, Lee SS, Seo DW, Lee SK, Kim MH, Han DJ, Kim SC, Lee JL. A randomised phase II study of modified FOLFIRI.3 vs modified FOLFOX as second-line therapy in patients with gemcitabine-refractory advanced pancreatic cancer. Br J Cancer. 2009 Nov 17;101(10):1658-63. doi: 10.1038/sj.bjc.6605374. Epub 2009 Oct 13. PMID 19826418
- See also: Yoo C et al. British Journal of Cancer 2009;101:1658-1663 — http://www.ncbi.nlm.nih.gov/pubmed/19826418